CLINICAL TRIAL: NCT02741544
Title: Revlimid® Capsules Special Drug Use-results Survey (in Patients With Newly-diagnosed Multiple Myeloma [NDMM])
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-Celgene-JP-PMS-003; U1111-1181-9845 (Registry Identifier: WHO)
Record Dates: First submitted 2016-04-05; First posted 2016-04-18 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: Second primary cancers; Cataracts; Newly-diagnosed multiple myeloma; Revlimid capsules
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Second Primary; Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with newly-diagnosed multiple myeloma (NDMM): Patients with newly-diagnosed multiple myeloma (NDMM) who are treated with Revlimid Capsules (Revlimid)

SUMMARY:
To understand the safety and efficacy of Revlimid® 2.5mg and 5 mg Capsules (hereinafter referred to as Revlimid) in all patients who are treated with it under the actual condition of use pursuant to the conditions of approval.

1. Planned registration period This period started on the date of initial marketing of Revlimid and will end at the time when the planned number of patients to be enrolled is reached.
2. Planned surveillance period This period started on the date of initial marketing of Revlimid and will end on the day when the approval condition related to all-case surveillance is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed multiple myeloma who are treated with Revlimid Capsules

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients with newly-diagnosed multiple myeloma (hereinafter referred to as "NDMM") who are treated with Revlimid Capsules (hereinafter referred to as "Revlimid", used by both 2.5 mg and 5 mg capsules).
Sampling Method: Probability Sample
Enrollment: 578 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 6 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Shinko Hospital, Kobe, Hyōgo, Japan